CLINICAL TRIAL: NCT03842020
Title: Population Pharmacokinetics and Pharmacodynamics of Amiodarone in Children": PK-AMIO
Brief Title: Pharmacokinetics of Amiodarone in Children
Acronym: PK-AMIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP180299; 2018-A02327-48 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2021-03

CONDITIONS: Heart Rhythm Disorder
Keywords: heart rhythm disorder; Amiodarone; Cardiac arrhythmias; Pediatric; Population pharmacokinetic (Pop PK); Modeling
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Amiodarone dosage (Experimental): Blood pharmacokinetics samples
  Interventions: Other: Blood pharmacokinetic samples

INTERVENTIONS:
Other: Blood pharmacokinetic samples — 1 or 3 sample(s) will be taken in the following time windows: [H0-H3]; [H5-H9] and just before the next set [H24], depending if the child is or is not admitted to hospital
  Other Names: Amiodarone dosage

SUMMARY:
PK-AMIO study is a population pharmacokinetic study of Amiodarone in children in order to :

* study the pharmacokinetic parameters (Pop PK) of Amiodarone in children;
* identify covariates explaining the variability of these pharmacokinetic parameters;
* study the relationship between the concentration, the efficacy of treatment and its tolerance to optimize the use of Amiodarone in pediatrics.

Indeed, there is no consensus on the optimal oral dosage in children. Few pharmacokinetic studies have been performed with only a small number of patients per study. Our study will include 70 children aged 0 to 18 years old.

DETAILED DESCRIPTION:
The incidence of supraventricular rhythm disorders in children is 1/250 to 1/1000. Amiodarone is used until the age of 1 year to limit the risk of recurrence. Efficiency is around 60% with no predictive factors identified. According to the study by Dallefeld (2018), unexplained inter-individual variability in pharmacokinetic parameters is 200%. Its adverse effects are numerous and affect 10% of patients. The concentration-effect relationship is poorly known. Amiodarone can cause hypotension and bradycardia. Liver and thyroid function should be monitored as well. Amiodarone is metabolised by cytochromes, mainly CYP3A4. Drug interactions and cytochrome variation in the neonatal period may alter its elimination kinetics. Pharmacokinetic studies have been conducted in adults with target concentrations of 0.5 to 2.5 mg/l.

The efficacy of oral amiodarone in children has been shown in studies in 1980; however, there is no consensus on optimal dosage. Despite its widespread use in children, few pharmacokinetic studies have been conducted in a small number of patients at different doses. The population pharmacokinetics and pharmacodynamics of Amiodarone in children, as well as its general and scientific interest, will be studied in this study. The lack of efficacy and the occurrence of adverse events of Amiodarone in children may be related to the large inter-individual pharmacokinetic variability.

Currently, more than 200 children treated with Amiodarone are being followed at Necker-Enfants malades Hospital.

This prospective study will be conducted in three paediatric services of Necker-Enfants malades Hospital in Paris, France.

Patient selection will take place in the 3 paediatric services. The senior physician proposes the study to holders of parental authority whose child receives or will receive the treatment during its follow-up or hospitalization.

After verification of the inclusion and exclusion criteria, the consent of the parents or parental authority and the child, according to his age, will be obtained.

After agreement, and/or signature of the parents and the non-oral opposition of the child in age to understand the information, the child is sampled according to the following scheme:

* The samples taken during the introduction of the treatment in hospital will be made to observe the pharmacokinetics at the first dose: 3 samples will be taken in the following time windows: [H0-H3]; [H5-H9] and just before the next dose administration (H24).
* During the maintenance treatment, a sample will be taken during a scheduled consultation or during a hospitalization.
* Blood PK samples will be drawn until 1 month after end of treatment.

All patients' samples will be kept for to be analyzed at the Pharmacology department of the Cochin hospital.

No intervention or no charge will be made for this study.

This population pharmacokinetic study in children aims to analyze the concentration-effectiveness and concentration-tolerance relationship to optimize its use.

ELIGIBILITY:
Inclusion Criteria:

* All children from 0 to 18 years old treated with Amiodarone for any rhythm disorder, and followed to Necker-Enfants maladies hospital.

Exclusion Criteria:

* Absence of parental and / or child consent
* Known liver dysfunction

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Maximal Concentration (Cmax) of amiodarone | Hour 0 to Hour 24
Area under the plasma concentration versus time curve (AUC) of amiodarone | Hour 0 to Hour 24
Clearance of amiodarone | Hour 0 to Hour 24
Volume of distribution of amiodarone | Hour 0 to Hour 24
Half time of amiodarone | Hour 0 to Hour 24

SECONDARY OUTCOMES:
Rhythm disorder | Day 0
  to assess Efficacity - Detection of the rhythm disorder on an ECG or scope (during hospitalization or consultation), or an ECG holter: absence of rhythm disorders at the atrial, junctional or ventricular level Or oral report from parents of rhythm disorder between 2 consultations (palpitation, heart rate acceleration)
Altered liver function | At the beginning of Amiodarone treatment until through study completion, an average of 18 months
  to assess Tolerance - from blood tests or clinical follow-up : gammaglutamyl transferase (GGT) U/L , Alkaline Phosphatase (ALP) U/L, Alanine Transaminase (ALT) U/L Aspartate Transaminase (AST) U/L,Total / conjugated/ free bilirubin µmol/L
Thyroid Dysfunction | At the beginning of Amiodarone treatment until through study completion, an average of 18 months
  to assess Tolerance - from blood tests or clinical follow-up : (TSH µmol/l, Free Tri-iodothyronine (FT3) and Free Thyroxine (FT4) pmol/L)
QT and corrected QT duration | At the beginning of Amiodarone treatment until through study completion, an average of 18 months
  to assess Tolerance - QT and corrected QT duration in milliseconds with an ECG
Blood pressure : (PAS)/(PAD) (mmHg) | At the beginning of Amiodarone treatment until through study completion, an average of 18 months
  to assess Tolerance

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc TRELUYER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Damien BONNET, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Sylvain RENOLLEAU, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Amelia LEHNERT, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehnert A, Foissac F, Bouazza N, Urien S, Oualha M, Renolleau S, Barbanti C, Di Marzio A, Bonnet D, Abdalla S, Zheng Y, Treluyer JM. Amiodarone/N-desethylamiodarone population pharmacokinetics in paediatric patients. Br J Clin Pharmacol. 2022 Dec;88(12):5369-5377. doi: 10.1111/bcp.15458. Epub 2022 Jul 29. PMID 35816412
- [Background] Dallefeld SH, Atz AM, Yogev R, Sullivan JE, Al-Uzri A, Mendley SR, Laughon M, Hornik CP, Melloni C, Harper B, Lewandowski A, Mitchell J, Wu H, Green TP, Cohen-Wolkowiez M. A pharmacokinetic model for amiodarone in infants developed from an opportunistic sampling trial and published literature data. J Pharmacokinet Pharmacodyn. 2018 Jun;45(3):419-430. doi: 10.1007/s10928-018-9576-y. Epub 2018 Feb 12. PMID 29435949
- [Background] Garson A Jr, Gillette PC, McVey P, Hesslein PS, Porter CJ, Angell LK, Kaldis LC, Hittner HM. Amiodarone treatment of critical arrhythmias in children and young adults. J Am Coll Cardiol. 1984 Oct;4(4):749-55. doi: 10.1016/s0735-1097(84)80402-7. PMID 6384328
- [Background] Coumel P, Fidelle J. Amiodarone in the treatment of cardiac arrhythmias in children: one hundred thirty-five cases. Am Heart J. 1980 Dec;100(6 Pt 2):1063-9. doi: 10.1016/0002-8703(80)90214-8. PMID 7446409
- [Background] Bucknall CA, Keeton BR, Curry PV, Tynan MJ, Sutherland GR, Holt DW. Intravenous and oral amiodarone for arrhythmias in children. Br Heart J. 1986 Sep;56(3):278-84. doi: 10.1136/hrt.56.3.278. PMID 3756044
- [Background] Pollak PT, Bouillon T, Shafer SL. Population pharmacokinetics of long-term oral amiodarone therapy. Clin Pharmacol Ther. 2000 Jun;67(6):642-52. doi: 10.1067/mcp.2000.107047. PMID 10872646